CLINICAL TRIAL: NCT06436573
Title: Mitro-annular Disjunction in Cardiac Magnetic Resonance
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Esposito, Professor, IRCCS San Raffaele
Other Study IDs: MAD-SIRM
Record Dates: First submitted 2024-03-27; First posted 2024-05-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Mitral Valve Prolapse Syndrome; Arrhythmogenic Bileaflet Mitral Prolapse; Mitral Valve Disorder
Keywords: Mitral annular disjunction, mitral prolapse, arrhthymia
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective cohort: Consecutive adult patients (age ≥18 years-old), submitted to Cardiac Magnetic Resonance independently by the clinical suspicions in the first semester of 2019 (from January to June 2019) that have signed an Informed Consent authorizing data collection for future retrospective clinical research protocols.
  Timelapse has been chosen to avoid the impact of COVID-19 pandemic.

SUMMARY:
Mitral annular disjunction (MAD) is an abnormal atrial displacement of the mitral valve leaflet hinge point. MAD is gaining clinical importance for several studies reporting its association to mitral valve prolapse (MVP), complex ventricular arrhythmias and sudden cardiac death.

On the other hand, other studies found MAD as an extremely diffuse anatomical variant of mitral valve annulus without any pathological implication.

Cardiac Magnetic Resonance is the non-invasive gold standard for myocardial characterization, with the possibility of accurate anatomical and functional evaluation associated to the evaluation of focal and interstitial fibrosis, resulting useful in the identification of arrhythmic substrate and for patients risk stratification. Additionally, Cardiac Magnetic Resonance (CMR) was found to be superior to echocardiography not only in term of tissue characterization, but also in the identification of small MAD.

Therefore, in relation to the scarcity of data about MAD prevalence and pathological potential, we set a large multicenter retrospective study aimed to evaluate prevalence of MAD in patients submitted to CMR independently by the clinical suspicion, and to evaluate the association with prolapse and arrhythmias.

DETAILED DESCRIPTION:
Multicenter retrospective study. All cardiac MRI study obtained during the first semester of 2019 will be screened in order to identify the presence and severity of MAD, it association to other myocardial condition such as bileaflet mitral valve prolapse, miltral regurgitation, curling, and focal and interstitial fibrosis at LGE and ECV evaluation.

Finally, the association between MAD and arrhythmias will be investigated.

ELIGIBILITY:
Inclusion Criteria:

• Consecutive adult patients (age ≥18 years-old), submitted to Cardiac Magnetic Resonance independently by the clinical suspicions in the first 6 month of 2019 (from January to June 2019) that have signed an Informed Consent authorizing data collection for future retrospective clinical research protocols

Exclusion Criteria:

• Pediatric patients (age <18 years-old), cardiac devices (implantable devices), previous mitral valve surgery, lack of LGE images, lack of clinical information about presence of arrhythmias. The timeline was selected to avoid the impact of COVID-19 pandemic on CMR availability, scheduling, and findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (age ≥18 years-old), submitted to Cardiac Magnetic Resonance independently by the clinical suspicions in the first semesterof 2019 (from January to June 2019)
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
the outcome will be the presence of MAD | 1 year
  The main objective of the present study is to investigate the prevalence of MAD in a large population undergoing CMR independently by the clinical suspicion. Therefore, the endpoint will be the prevalence of MAD in the examined population and the outcome will be the presence of MAD.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Esposito, MD, Principal Investigator — IRCCS San Raffaele Institute
Locations (1):
- IRCCS San Raffaele, Milan, Italy

REFERENCES:
- [Background] Kulkarni AA, Chudgar PD, Burkule NJ, Kamat NV. Mitral Annulus Disjunction and Arrhythmic Mitral Valve Prolapse: Emerging Role of Cardiac Magnetic Resonance Imaging in the Workup. Indian J Radiol Imaging. 2022 Aug 30;32(4):576-581. doi: 10.1055/s-0042-1754357. eCollection 2022 Dec. PMID 36451946
- [Background] Bennett S, Thamman R, Griffiths T, Oxley C, Khan JN, Phan T, Patwala A, Heatlie G, Kwok CS. Mitral annular disjunction: A systematic review of the literature. Echocardiography. 2019 Aug;36(8):1549-1558. doi: 10.1111/echo.14437. Epub 2019 Aug 5. PMID 31385360
- [Background] Chess RJ, Mazur W, Palmer C. Stop the Madness: Mitral Annular Disjunction. CASE (Phila). 2023 Jan 18;7(3):116-118. doi: 10.1016/j.case.2022.12.004. eCollection 2023 Mar. PMID 37065832
- [Background] Faletra FF, Leo LA, Paiocchi VL, Schlossbauer SA, Pavon AG, Ho SY, Maisano F. Morphology of Mitral Annular Disjunction in Mitral Valve Prolapse. J Am Soc Echocardiogr. 2022 Feb;35(2):176-186. doi: 10.1016/j.echo.2021.09.002. Epub 2021 Sep 8. PMID 34508838
- [Background] Bennett S, Tafuro J, Duckett S, Appaji A, Khan JN, Heatlie G, Cubukcu A, Kwok CS. Definition, prevalence, and clinical significance of mitral annular disjunction in different patient cohorts: A systematic review. Echocardiography. 2022 Mar;39(3):514-523. doi: 10.1111/echo.15299. Epub 2022 Feb 4. PMID 35122307
- [Background] Dejgaard LA, Skjolsvik ET, Lie OH, Ribe M, Stokke MK, Hegbom F, Scheirlynck ES, Gjertsen E, Andresen K, Helle-Valle TM, Hopp E, Edvardsen T, Haugaa KH. The Mitral Annulus Disjunction Arrhythmic Syndrome. J Am Coll Cardiol. 2018 Oct 2;72(14):1600-1609. doi: 10.1016/j.jacc.2018.07.070. PMID 30261961